CLINICAL TRIAL: NCT01510132
Title: Post Marketing Surveillance Study to Evaluate the Safety Profile of Travacom (Travoprost/Timolol Fixed Combination) in Patients With Open-Angle Glaucoma or Ocular Hypertension Across India
Brief Title: Travacom Post Marketing Surveillance Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-11-012
Record Dates: First submitted 2012-01-11; First posted 2012-01-13 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Travacom (Experimental): Travoprost/timolol fixed combination self-administered at the rate of 1 drop per eye, one time a day, at approximately 8 a.m. each day for 8 weeks.
  Interventions: Drug: Travoprost/timolol fixed combination (Travacom)

INTERVENTIONS:
Drug: Travoprost/timolol fixed combination (Travacom) — Commercially-marketed drug for the treatment of open-angle glaucoma or ocular hypertension
  Other Names: Travacom

SUMMARY:
The purpose of this multi-center, open label, single arm, post-marketing surveillance study is to assess the safety of Travacom in patients with open-angle glaucoma or ocular hypertension who are insufficiently responsive to beta-blockers, prostaglandins, or other intraocular pressure-lowering (IOP) medication and when use of Travacom is considered appropriate.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Open-angle glaucoma or ocular hypertension insufficiently responsive to betablockers, prostaglandins, or other intraocular pressure-lowering (IOP) agents and when the use of Travacom is considered appropriate.
* Discontinued use of all other ocular hypotensive medications prior to receiving the study medication for the entire course of the study.
* Mean IOP not greater than 36 mmHG in either eye.
* Read, sign, and date (or legal representative) the Informed Consent prior to the start of any study-related procedures.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential (not postmenopausal for at least one year or not surgically sterile) who are currently pregnant, have a positive result on the urine pregnancy test at Screening, intend to become pregnant during the study period, are breastfeeding, or do not agree to use an adequate birth control method to prevent pregnancy throughout the study.
* Chronic, recurrent, or severe inflammatory eye disease, such as scleritis, uveitis, or herpes keratitis.
* History of clinically significant or progressive retinal disease.
* Best corrected visual acuity (BCVA) score worse than 20/80 Snellen.
* Bronchial asthma or related history that would preclude safe administration of a topical beta-blocker.
* Severe, unstable, or uncontrolled cardiovascular, hepatic, or renal disease or related history that would preclude safe administration of a topical beta-adrenergic blocking agent.
* History of spontaneous or current hypoglycemia or uncontrolled diabetes.
* Known medical allergy, hypersensitivity, or poor tolerance to any component of Travacom deemed clinically significant in the opinion of the Principal Investigator.
* Use of any additional topical or system ocular hypotensive medication during the study.
* Participation in any other investigational study within 30 days prior to Screening visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Extent of exposure | Up to 8 weeks
  Extent of exposure is calculated as days on therapy. Days on therapy is defined as the difference in days between the date of exit (last) instillation as recorded on the last visit and the visit at which medication was first administered.
Adverse events | Up to 8 weeks
  Any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. Adverse events will be collected spontaneously and systematically at each scheduled study visit and may be collected at any unscheduled visit that occurs during the study. Adverse events will be documented on Adverse Events Forms and will be reported by MedDRA preferred terminology.